CLINICAL TRIAL: NCT02259322
Title: Treatment of Loss of Control Eating Following Bariatric Surgery
Brief Title: Loss of Control Eating Following Weight Loss Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1205010224; R01DK098492-01A1 (NIH)
Record Dates: First submitted 2014-09-29; First posted 2014-10-08 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Loss of Control Eating
Keywords: Bariatric surgery; Weight loss surgery; Behavioral weight loss treatment; Cognitive behavioral therapy; Behavioral treatment; Obesity; Morbid obesity; Binge eating; Binge eating disorder; Loss of control eating; Overeating
MeSH Terms: conditions — Obesity; Obesity, Morbid; Bulimia; Binge-Eating Disorder; Hyperphagia | interventions — Standard of Care; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Standard-of-Care (Active Comparator): Standard-of-care is the continuation of any treatment or recommendations participants receive from his/her bariatric surgeon/team.
  Interventions: Behavioral: Standard-of-Care
- Behavioral Weight Loss Treatment (Experimental): Guided self-help Behavioral Weight Loss Treatment
  Interventions: Behavioral: Behavioral Weight Loss Treatment
- Cognitive Behavioral Therapy (Experimental): Guided self-help Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Standard-of-Care — Standard-of-Care with bariatric team. Participants will be encouraged to continue their care with their bariatric team.
  Arms: Standard-of-Care
Behavioral: Behavioral Weight Loss Treatment — Biweekly individual guided self-help sessions for 3 months
  Arms: Behavioral Weight Loss Treatment
Behavioral: Cognitive Behavioral Therapy — Biweekly individual guided self-help sessions for 3 months
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study will test the effectiveness of two distinct behavioral treatments for loss of control eating following bariatric surgery:

1. Behavioral Weight Loss Treatment
2. Cognitive Behavioral Therapy

These treatments will be compared to Standard-of-Care.

ELIGIBILITY:
Inclusion Criteria:

* Gastric bypass surgery or sleeve gastrectomy patients from Yale Bariatric/Gastrointestinal Surgery Program
* 5-8 months post-bariatric surgery
* Regular loss of control eating (once weekly during past month)
* Read English proficiently enough to read patient self-care materials and study assessments
* Available for duration of treatment plus follow-up period
* Agree to study procedures

Exclusion Criteria:

* Current enrollment in a formal exercise program
* Medical status judged by the surgeon as contraindication (rare instances of need for additional surgery or medical instability)
* Unable to ambulate
* Current medications that influence eating/weight
* Current substance dependence or other severe psychiatric disturbance (e.g., suicidality) that requires immediate treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Loss of Control Eating Frequency (Categorical) | Post-treatment (at 3 months)
  Loss of Control eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency is defined categorically (presence or absence of loss of control eating).
Loss of Control Eating Frequency (Categorical) | 24 month follow-up (an average of 24 months following treatment)
  Loss of Control eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency is defined categorically (presence or absence of loss of control eating).
Loss of Control Eating Frequency (Continuous) | Post-treatment (at 3 months)
  Loss of Control eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency also is defined continuously (analyzed dimensionally).
Loss of Control Eating Frequency (Continuous) | 24 month follow-up (an average of 24 months following treatment)
  Loss of Control eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency also is defined continuously (analyzed dimensionally).
Body Mass Index (BMI) | Post-treatment (at 3 months)
  BMI is calculated using measured height and weight.
Body Mass Index (BMI) | 24 month follow-up (an average of 24 months following treatment)
  BMI is calculated using measured height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, Ph.D., Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Lawson JL, Wiedemann AA, Carr MM, Ivezaj V, Duffy AJ, Grilo CM. Examining Sleep Quality Following Sleeve Gastrectomy Among Patients with Loss-of-Control Eating. Obes Surg. 2019 Oct;29(10):3264-3270. doi: 10.1007/s11695-019-03981-7. PMID 31197602